CLINICAL TRIAL: NCT05413538
Title: Effects of a Mindfulness-Based Intervention Delivered Via Instant Messaging on Parents' Wellbeing: A Randomized Controlled Trial and Investigation of Moderators
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lam Lun Wai Doris, Principal Investigator, Graduate Student in Clinical Psychology, Department of Psychology, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBRE(R)-21-039
Record Dates: First submitted 2022-06-04; First posted 2022-06-10 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Parents; Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will be invited to listen to a 15-minute mindfulness instructional recording delivered daily through an instant messaging application and to practice accordingly for 14 consecutive days at their own choice of time and place.
  Interventions: Behavioral: Mindfulness training
- Waitlist control group (No Intervention): The waitlist control group will only be required to complete the demographic information, pre, post experiment and follow-up questionnaires before they receive the mindfulness training intervention.

INTERVENTIONS:
Behavioral: Mindfulness training — The intervention recordings will teach the basic concepts of mindfulness through simple guided meditations with content supported by science. Each recording has the same format that included (1) a daily theme, (2) a meditation exercise echoing the theme, (3) a suggested exercise for practice, and (4) an invitation for participants to give a short response to their meditation experience at the end of the recording.
  Arms: Experimental Group

SUMMARY:
This research investigates the effects of mindfulness practice on mental wellbeing with the instruction recordings delivered via existing instant messaging applications, Whatsapp. The two-week mindfulness program targets parents with children in Secondary School or below. This research also explores how parenting and attachment styles moderate the intervention effects.

ELIGIBILITY:
Inclusion Criteria:

Parents with at least one child who is in Secondary School or below

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-09-28 (Estimated); Study Completion 2022-09-28 (Estimated)

PRIMARY OUTCOMES:
Parental Stress Scale | Change from Baseline Parental Stress Scale at immediately after the intervention and two weeks after intervention
  The Parental Stress Scale was used to measure self-perceived stress specific to the parenting role. Parental Stress Scale was originally developed by Berry and Jones (1995) to measure parental feelings and experiences in terms of rewards, satisfaction, controllability, and stress. The minimum score was 0 and the maximum score was 64. A score of 0 represents lowest level of parental stress possible, whereas a score of 64 represents highest level of parental stress. Higher scores indicate worse outcome.
Interpersonal Mindfulness in Parenting Scale | Change from Baseline Interpersonal Mindfulness in Parenting scale at immediately after the intervention and two weeks after intervention
  The 31-item Interpersonal Mindfulness in Parenting scale was adopted to measure parents' self-reported engagement in mindful parenting (Duncan, 2007). The minimum score was 0 and the maximum score was 155. A score of 0 represents lowest level of parental mindfulness, whereas a score of 155 represents highest level of parental mindfulness possible. Higher scores indicate better outcome.
Non-attachment to Self Scale | Change from Baseline Non-attachment to Self Scale at immediately after the intervention and two weeks after intervention
  Non-attachment to Self Scale measures the absence of fixation on self-related concepts, thoughts and feelings, and a capacity to flexibly interact with these concepts, thoughts and feelings without trying to control them (Whitehead et al., 2018). The minimum score was 0 and the maximum was 49. The higher the score the more nonattached the participant. Higher scores indicate better outcome.
Nonattachment Scale - Short Form | Change from Baseline Nonattachment Scale - Short Form at immediately after the intervention and two weeks after intervention
  Nonattachment Scale measures an individual's release from mental fixations in a flexible, balanced way of relating to one's experiences without clinging to or suppressing them (Chio, Lai, & Mak, 2018). The minimum score was 0 and the maximum was 48. The higher the score the more nonattached the participant. Higher scores indicate better outcome.
Peace of mind | Change from Baseline Peace of mind Scale - Short Form at immediately after the intervention and two weeks after intervention
  Peace of mind scale measures an individual's internal state of peacefulness and harmony (Lee et al., 2013).The minimum score was 0 and the maximum score was 35. Higher scores reflect higher levels of peace of mind. Higher scores indicate better outcome.

SECONDARY OUTCOMES:
The Experiences in Close Relationship Scale-Short Form | Change from Baseline The Experiences in Close Relationship Scale - Short Form at immediately after the intervention and two weeks after intervention
  The Experience in Close Relationship Scale is a 12 item self-report adult attachment style questionnaire focused on close relationships (Brennan, Clark & Shaver, 1998). It provides data on two continuous scales concerning the extent to which participants show attachment dimensions: anxiety and avoidance. The scale consists of 12 items which participants respond to on a seven-point scale. The minimum score was 0 and the maximum score for each scale was 72. The lower the score the more securely attached the participant. Higher scores indicate worse outcome.
Training Scale | Change from Baseline Training Scale at immediately after the intervention and two weeks after intervention
  The Training Scale measures child-rearing items specific to the Chinese culture (Chao, 1994). The training scale covered two areas, "ideologies on child development and learning" (involving seven items) and "ideologies on the mother-child relationship" (involving six items). The minimum score was 0 and the maximum score was 65. The higher the score the more the participant pertains to chiao shun, or training.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No